CLINICAL TRIAL: NCT02088593
Title: The Effect of Improving Sleep and Circadian Rhythms on Affective Symptoms In First Year Medical Students
Brief Title: Simulated Dawn Med Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: University at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dawn
Record Dates: First submitted 2014-02-26; First posted 2014-03-17 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Depression; Anxiety; Fatigue; Sleepiness; Sleep Disruption
Keywords: Medical Students
MeSH Terms: conditions — Depression; Anxiety Disorders; Fatigue; Sleepiness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAWN simulation (Experimental): Simulated Dawn Light box
  Interventions: Device: Simulated Dawn Light Box; Behavioral: Sleep Hygiene instructions
- Sleep hygiene instructions read aloud (Active Comparator): Standard sleep hygiene instructions were read aloud.
  Interventions: Behavioral: Sleep Hygiene instructions

INTERVENTIONS:
Device: Simulated Dawn Light Box — per3 model of Naturebright It was set at the participants habitual wake time, and automatically began ramping between 30 and 90 minutes prior to that time (based upon participant preference). The ramp increased in a curvilinear fashion, mimicking sunrise during the summer at 45 degrees North latitude and reached a maximum light intensity of 300lux. They were allowed to switch the lamp off during the ramp period, and sleep in on off days, but were asked to allow the light to begin its ramp.
  Other Names: per3 model of Naturebright
  Arms: DAWN simulation
Behavioral: Sleep Hygiene instructions — Sleep Hygiene instructions read aloud

SUMMARY:
Medical students score higher than the general population on measures of depression, anxiety, fatigue, poor sleep and sleepiness. Data suggest that disparages in circadian phase might contribute to these problems. From an internal validity standpoint, first year medical students are an ideal group to study. The majority of the students will be matched on variables such as education, age, and intelligence. However, more importantly, they have a nearly identical life style when it comes to factors such as schedule, living conditions, level of stress, and timing of stressors. The specific aim and hypothesis is:Medical students randomized to sleep hygiene counseling plus simulated dawn will report less depression, anxiety, fatigue, sleepiness, and sleep disruption (as measured by standardized questionnaires) than students randomized to just sleep hygiene counseling.

DETAILED DESCRIPTION:
There is a substantial and growing body of literature that has identified medical students as a group that suffers from increased levels of depression, anxiety, and other markers of "psychological distress". Other studies have demonstrated that in conjunction with the "psychological distress", medical students suffer from sleep deprivation, sleep disruption, and daytime sleepiness. Finally there is some preliminary evidence that residents and interns show increased symptoms of fatigue. It might reasonably be assumed that all of these symptoms are inter-related and more importantly detrimental to both the student and those patients under their care. There have been interventional studies aimed at educating participants on stress management, however these attempts have had only limited success.

Circadian rhythms are biological rhythms that contribute to most of our bodies' physiological processes. It has been determined that light is the major environmental cue that influences the setting of our circadian rhythm. Under ideal circumstances exposure to natural sunlight is sufficient to maintain a consistent and synchronized circadian rhythm. Often times this is not the case. Reduced exposure to natural light and increased exposure to artificial light are just two influencing factors.

Artificial light therapy has been successfully applied to the treatment of disorders of circadian rhythms as well as the treatment of some affective disorders. Most notably, light therapy has been shown to be effective in treating symptoms of depression and sleep disruption, specifically in patients with seasonal affective disorder, non-seasonal major depression, delayed sleep phase syndrome, advanced sleep phase syndrome, and sub-syndromal levels of each of these.

The theoretical mechanism of action is reviewed by Terman et al and asserts that morning bright light therapy advances and stabilizes the circadian rhythm of individuals who have delayed or drifting rhythms. There is subsequent synchronization and entrainment of the individual's endogenous rhythm with the environmental rhythm of daily life as reviewed in.

The timing, duration, and type of light delivered are of paramount concern, as improper delivery of therapy has been shown to have no advantage over placebo. One method of light delivery is simulated dawn light therapy. Simulated dawn light therapy works by gradually increasing light exposure over a specified period of time at the end of the sleep period. This gradually increasing light exposure during the sleep period is in contrast to traditional light therapy, which is delivered at full intensity after wake time. Simulated dawn has shown great promise as being just as effective as traditional light therapy but with the additional advantages of being more time efficient, easier to use, and more easily tolerated. All of these factors are important considerations in the application of this intervention to medical students, as being short on time and under significant stress are both hallmarks of medical education. The following proposal is a novel approach, using light therapy, to improve the mental well-being of first year medical students.

ELIGIBILITY:
Inclusion Criteria:

* Being a first year medical student
* Good academic standing after the first module
* Reporting attending morning lectures regularly.

Exclusion Criteria:

* No reported history of psychiatric illness,sleep illness, ophthalmic illness
* No current use of photosensitizing medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Sleep quality | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- University at Buffalo, Buffalo, New York, United States